CLINICAL TRIAL: NCT00524914
Title: Apomorphine Effect on Nociceptive Perception in Parkinson's: a Clinical and Imaging Study.
Acronym: APODOUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: LLAU Marie-Elise, University Hospital Toulouse
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0602308; PHRC 2006
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Pain; Nociceptive threshold; Functional imaging; Cerebral activity; Dopamine agonist.
MeSH Terms: conditions — Parkinson Disease; Pain | interventions — Apomorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Apomorphine
  Interventions: Drug: apomorphine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: apomorphine — Acute apomorphine subcutaneous 3 mg
  Arms: 1
Drug: placebo — placebo subcutaneous
  Arms: 2

SUMMARY:
Patients suffering from Parkinson's disease (PD) frequently experienced painful sensations. We suppose that painful symptoms could be related to the neurotransmitter deficit of PD. So, we would like to evaluate the involvement of dopaminergic system in nociceptive processing in PD patients. The objectives of this study is to assess and to compare the effect of a dopamine agonist administration on the nociceptive threshold and on the cerebral activity using positrons emission tomography (PET scan) in two groups of PD patients (in 16 painful PD patients and in 16 pain free PD patients). We hypothesise that dopamine agonist could normalise nociceptive threshold and cerebral activity which were both abnormal in PD patients. Moreover, we think that painful PD patients could be more improved by dopamine agonist than pain free PD patients.

DETAILED DESCRIPTION:
Patients suffering from Parkinson's disease (PD) frequently experienced painful sensations. Painful complaints with various description (muscle cramps, painful dystonia, aching, numbness, tingling, burning, vibrating, lancinating) are described and can or cannot be related to motor symptoms. Physiopathology of pain in PD is discussed. It has been suggested that the occurrence of painful symptoms could be in part due to central modification of nociception and basal ganglia damage and the dopaminergic deficit would be expected to eliminate the inhibitory influence on thalamic nociceptive activity. Recently, data have shown that PD patient had a lower nociceptive threshold than healthy volunteers. Our team has reported that levodopa administration normalised this nociceptive threshold and decreased cerebral activity measured with positrons emission tomography (PET- H215O during experimental nociceptive stimulation) in several nociceptive cortical areas which were overactive in PD. These findings suggest that central dopamine system plays an important part in the control of the nociceptive pathways in PD. Nevertheless, in the central nervous system, levodopa could be converted in dopamine but also in noradrenaline modulating noradrenergic system. In order to confirm the involvement of dopaminergic system in nociceptive processing in PD, we would like to assess a specific drug of dopamine system (a dopamine agonist, apomorphine) in PD patients.

The primary objective of this study is to assess the effect of dopamine agonist acute administration versus placebo on the nociceptive subjective threshold in two groups of PD patients (painful PD patients, n =16 and pain free PD patients, n = 16). This is a controlled cross over, double blind, randomised study.

The secondary objectives are to assess and to compare the apomorphine effect on the objective nociceptive threshold (nociceptive flexion reflex) and on the activation of cerebral areas using functional imaging (TEP- H215O) during experimental nociceptive stimulation in the two groups of PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Parkinson's disease
* PD patients with a Hoehn et Yahr < à 3 (Hoehn et Yahr 1967)
* PD patients treated by dopaminergic drugs (levodopa, dopamine agonist, IMAO-B, ICOMT…)
* Painful PD patients : PD patients suffering from chronic pain (> 3 months) which is related to PD and suggests neuropathic pain
* Pain free PD patients : PD patients without any pain related to PD.

Exclusion Criteria:

* Patients with chronic disease resulting in chronic pain (severe arthosis….)
* PD patients with a Hoehn et Yahr stage > 3 (Hoehn et Yahr 1967)
* Patients with cancer
* Patients who underwent a PET scan in the last three months
* Pregnancy
* Patients with a contra indication of use of apomorphine or domperidone.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is subjective nociceptive threshold using thermotest. We determinate thermal nociceptive threshold using a Peltier- based contact temperature stimulation device with a contact thermode. | the primary outcome is measured after acute administration of apomorphine ( after 30 minutes )

SECONDARY OUTCOMES:
Objective nociceptive threshold using the nociceptive flexion reflex (RIII) which can be elicited by a nociceptive electrical stimulation to the sural nerve and recorded in the ipsilateral Biceps Femoris muscle. | after acute administration of apomorphine
Cerebral activity using H215O PET analysis of regional Cerebral Blood Flow (rCBF) on subjects while they received alternate randomized noxious (defined as pain threshold) and innocuous stimuli. | After administration of apomorphine

CONTACTS AND LOCATIONS:
Overall Officials: Christine BREFEL-COURBON, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service de Neurologie, Toulouse, Toulouse, France